CLINICAL TRIAL: NCT06496958
Title: CO2 Insufflation Colonoscopy with an Abdominal Compression Device and Water Exchange Colonoscopy to Reduce Manual Assistance by Endoscopy Staff: a Multicenter Randomized Trial
Brief Title: Water Exchange and CO2 Insufflation with Abdominal Compression Device to Reduce Manual Assistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Collaborators: E-Da Dachange Hospital, Kaohsiung, Taiwan (Unknown); The Sepulveda Ambulatory Care Center, VAGLAHS, UCLA in the USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EGH-2024
Record Dates: First submitted 2024-06-20; First posted 2024-07-11 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Manual Pressure; Repositioning; Colonoscopy; Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CO2 insufflation colonoscopy with an abdominal compression device (Experimental): Colonoscopic insertion will be performed with CO2 insufflation with assistance by an abdominal compression device.
  Interventions: Device: CO2 insufflation with an abdominal compression device
- CO2 insufflation colonoscopy with a sham abdominal compression device (Sham Comparator): Colonoscopic insertion will be performed with CO2 insufflation in standard method. A sham abdominal compression device will be used as a sham comparator.
  Interventions: Device: CO2 insufflation with a sham abdominal compression device
- Water exchange colonoscopy (Active Comparator): Colonoscopic insertion will be performed with water exchange method.
  Interventions: Device: Water exchange colonoscopy

INTERVENTIONS:
Device: CO2 insufflation with an abdominal compression device — For participants randomized to the intervention group, the back brace support belt, Maxbelt (me3 type, Nippon Sigmax Co., Tokyo, Japan), will be applied around the circumference of the lower abdomen. Five sizes of Maxbelt will be employed in this study. According to the manufacturer, the ultra small-size (XS-size) belt will be used in those patients with an abdominal circumference of 55 cm-65 cm, the small-size (S-size) belt will be used in those patients with an abdominal circumference of 65 cm-75 cm, the medium-size (M-size) belt will be used for a circumference of 75 cm-85 cm, the large-size (L-size) belt will be used for a circumference of 85 cm-95 cm, and the ultra large-size (XL-size) will be used for a circumference of 95 cm-105 cm. Once applied, participants will be asked to assess and confirm that the belt is fastened tightly but not uncomfortably.
  Arms: CO2 insufflation colonoscopy with an abdominal compression device
Device: CO2 insufflation with a sham abdominal compression device — The study coordinator will fit the sham device in a private bay alone with the patient. For participants randomized to the sham control group, a larger-sized Maxbelt with loose fitting will be used as a sham device. The L-size Maxbelt will be used in those patients with an abdominal circumference of 55 cm-71 cm, the XL-size Maxbelt will be used in in those patients with an abdominal circumference of 72 cm-88 cm, and the 2 XL-size Maxbelt will be used in in those patients with abdominal circumference 89 cm-105 cm.
  Arms: CO2 insufflation colonoscopy with a sham abdominal compression device
Device: Water exchange colonoscopy — In those patients assigned to the water exchange (WE) group, the air pump will be turned off during the insertion phase of colonoscopy, while the colon is irrigated with warm-to-touch distilled water or half normal saline using a flushing pump. The WE approach involves the simultaneous infusion of water to facilitate luminal expansion and suction of unclean water during insertion. Any encountered air pockets will be aspirated to ensure optimal WE maneuvers in salvage cleaning.
  Arms: Water exchange colonoscopy

SUMMARY:
The goal of this trial is to evaluate whether water exchange colonoscopy and CO2-insufflation colonoscopy with an abdominal compression device (Maxbelt me3 type, Nippon Sigmax Co., Tokyo, Japan) can achieve a significantly lower proportion of patients requiring manual abdominal pressure during colonoscopic insertion compared with CO2 insufflation alone.

DETAILED DESCRIPTION:
This will be a three-arm multicenter parallel randomized controlled trial (RCT) designed to compare the frequency of ancillary manual assistance (abdominal pressure and/or position change) between CO2-insufflation colonoscopy with Maxbelt (intervention group), CO2-insufflation colonoscopy with sham device (sham control group), and water exchange (WE) colonoscopy (WE group). Enrolled patients will be randomized in a 1:1:1 ratio to either the intervention, sham control, or WE group. This will be a comparison of three different methods (CO2 with interventional device, CO2 with sham device, WE) to see which one is better at decreasing the need for manual assistance by endoscopy staff during colonoscopic insertion.

This study will be conducted in two hospitals in Taiwan: Evergreen General Hospital at Taoyuan and E-Da Dachange Hospital at Kaohsiung. The Sepulveda Ambulatory Care Center, VAGLAHS, UCLA in the USA will be a non-recruiting participating site. This planned RCT will span 30 months (from June 2024 to November 2026), including 3 months for the initial setup and 3 months for the final analysis. The study site possesses state-of-the-art colonoscopy equipment setups, and the investigators are WE colonoscopy research experts.

Patients aged 45-75 y/o at average risk of colorectal cancer who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site, stratified by investigator and type of colonoscopy (screening, surveillance, or positive fecal immunochemical test result). Mode of sedation will include conscious sedation (fentanyl plus midazolam) or full sedation (propofol with fentanyl plus midazolam) . Randomization will be carried out by computer-generated sequences using a block design (four participants per block).

CO2 with interventional device group: The Maxbelt will be applied around the circumference of the lower abdomen just below the umbilicus based on patient's abdominal circumference. Five sizes of Maxbelt will be employed in this study: XS-size for 55-65 cm circumference, S-size for 65-75 cm circumference, M-size for 75-85 cm circumference, L-size for 85-95 cm circumference, and XL-size for 95-105 cm circumference. Once applied, participants will be asked to assess and confirm that the belt is fastened tightly but not uncomfortably.

CO2 with sham device group: A two-size larger Maxbelt with loose fitting will be used as a sham device: L-size will be used for 55-71 cm circumference, XL-size will be used for 72-88 cm circumference, and 2 XL-size will be used for 89-105 cm circumference.

WE group: The air pump will be turned off during the insertion phase of colonoscopy, while the colon is irrigated with warm-to-touch distilled water or half normal saline using a flushing pump. The WE approach involves the simultaneous infusion of water to facilitate luminal expansion and suction of unclean water during insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-80 years having an average risk for colorectal cancer who plan to undergo sedated outpatient colonoscopy for screening, surveillance, and those who have received a positive fecal immunochemical test result

Exclusion Criteria:

* Patients with hereditary colorectal cancer syndrome, including familial adenomatous polyposis and hereditary nonpolyposis colorectal cancer (Lynch syndrome)
* Patients with serrated polyposis syndrome
* Patients with known or suspected inflammatory bowel disease
* Patients with a history of colorectal cancer or other intra-abdominal malignancy
* Patients with a history of colorectal resection
* Patients with a history of abdominal aortic aneurysm, cirrhosis, ascites, or other severe comorbid illnesses
* Patients with recent wounds or skin rash on the anterior abdominal wall and back
* Patients with known ventral hernia
* Patients with unsedated procedure
* Patients with planned bidirectional endoscopy
* Patients with body mass index >35 kg/m2
* Patients with waist circumference <55 cm or >105 cm
* Patients with known or suspected gastroparesis
* Patients with planned therapeutic procedures (e.g., hemostasis, removal of a large polyp)
* Patients with mental retardation
* Pregnant women or those planning pregnancy
* Patients unwilling to participate in the study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of manual pressure | One day
  The proportion of patients who need at least one application of manual abdominal pressure during colonoscopic insertion.

SECONDARY OUTCOMES:
Frequency of repositioning | One day
  The proportion of patients who need at least one application of position change during colonoscopic insertion.
Ergonomic pain of after colonoscopy | One day
  The musculoskeletal pain experienced by the assisting nurse will be reported based on a 5-point visual analogue scale score immediately after a procedure by using a questionnaire.
Colonoscopy difficulty | One day
  The colonoscopy difficulty assessed by the endoscopist will be reported using a 5-point visual analogue scale score immediately after completion of the procedure by using a questionnaire.
Post-colonoscopy abdominal pain | One day
  The pain experienced by the patient will be recorded in the recovery room post-procedure via a questionnaire using a 5-point visual analogue scale score.
Cecal intubation time | One day
  The cecal intubation time is defined as the time spanning from anal insertion to colonoscopic intubation of cecum.
Withdrawal time | One day
  The withdrawal time is defined as the time spanning from cecal intubation to colonoscope withdrawal from the anus.
Adenoma detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  The proportion of patients with at least one conventional adenoma of any size.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Liang Cheng, Principal Investigator — Evergreen General Hospital
Locations (2):
- Taiwan (2):
  - E-Da Dachang Hospital, Kaohsiung City
  - Evergreen General Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crockett SD, Cirri HO, Kelapure R, Galanko JA, Martin CF, Dellon ES. Use of an Abdominal Compression Device in Colonoscopy: A Randomized, Sham-Controlled Trial. Clin Gastroenterol Hepatol. 2016 Jun;14(6):850-857.e3. doi: 10.1016/j.cgh.2015.12.039. Epub 2016 Jan 6. PMID 26767313
- [Background] Toyoshima O, Nishizawa T, Sakitani K, Yamakawa T, Yoshida S, Fukagawa K, Hata K, Ishihara S, Suzuki H. Colonoscopy using back brace support belt: A randomized, prospective trial. JGH Open. 2019 Nov 7;4(3):441-445. doi: 10.1002/jgh3.12276. eCollection 2020 Jun. PMID 32514451
- [Background] Costello B, James T, Hall C, Shergill A, Schlossberg N. Does Manual Abdominal Pressure During Colonoscopy Put Endoscopy Staff and Patients at Risk? Experiences of Endoscopy Nurses and Technicians. Gastroenterol Nurs. 2023 Sep-Oct 01;46(5):386-392. doi: 10.1097/SGA.0000000000000756. Epub 2023 Jun 8. PMID 37289853
- [Background] Crockett S, Dellon ES, Biggers L, Ernst DA. Use of Patient Abdominal Compression Device Reduces Staff Musculoskeletal Pain Associated With Supporting Colonoscopy: Results From a Randomized Controlled Trial. Gastroenterol Nurs. 2021 Mar-Apr 01;44(2):136-145. doi: 10.1097/SGA.0000000000000550. PMID 33795622
- [Background] Cadoni S, Falt P, Gallittu P, Liggi M, Mura D, Smajstrla V, Erriu M, Leung FW. Water Exchange Is the Least Painful Colonoscope Insertion Technique and Increases Completion of Unsedated Colonoscopy. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1972-80.e1-3. doi: 10.1016/j.cgh.2015.04.178. Epub 2015 May 5. PMID 25956838
- [Background] Hsieh YH, Tseng CW, Hu CT, Koo M, Leung FW. Prospective multicenter randomized controlled trial comparing adenoma detection rate in colonoscopy using water exchange, water immersion, and air insufflation. Gastrointest Endosc. 2017 Jul;86(1):192-201. doi: 10.1016/j.gie.2016.12.005. Epub 2016 Dec 15. PMID 27988288